CLINICAL TRIAL: NCT02787629
Title: Comparison of Simultaneous Endotracheal Tube Insertion With GlideScope Use: a Pilot Study
Brief Title: Comparison of Simultaneous Endotracheal Tube Insertion With GlideScope Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107322
Record Dates: First submitted 2016-05-25; First posted 2016-06-01 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Intubation; Videolaryngoscopy
Keywords: D007440

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simultaneous (Experimental): Simultaneous Intubation with GlideScope and ETT inserted simultaneously
  Interventions: Procedure: Simultaneous Intubation
- Control Standard (Active Comparator): Standard Intubation with GlideScope inserted first and ETT inserted after the GlideScope view is obtained
  Interventions: Procedure: Standard Intubation

INTERVENTIONS:
Procedure: Simultaneous Intubation — Intubation with GlideScope and ETT inserted simultaneously
  Arms: Simultaneous
Procedure: Standard Intubation — Intubation with GlideScope inserted first and ETT insertion after the GlideScope view is obtained
  Arms: Control Standard

SUMMARY:
Patients presenting for elective surgery requiring orotracheal intubation will be randomized to having the ETT inserted into the pharynx simultaneous to GlideScope insertion and then having the ETT advanced under GlideScope guidance into the trachea, or, being intubated in the more common fashion with the GlideScope being inserted first and having the ETT then advanced via the pharynx into the trachea.

DETAILED DESCRIPTION:
Patients presenting for elective surgery requiring orotracheal intubation will be randomized to having the ETT inserted into the pharynx simultaneous to GlideScope insertion and then having the ETT advanced under GlideScope guidance into the trachea, or, being intubated in the more common fashion with the GlideScope being inserted first and having the ETT then advanced via the pharynx into the trachea. The primary outcome is time to intubation. Secondary outcomes include: 1) Ease of intubation as noted by operator (measured on a 10-cm Visual Analogue Scale) 2) Number of intubation attempts 3) Number of failures to intubate 4) Use of external laryngeal pressure 5) Laryngoscopic grade distribution

ELIGIBILITY:
Inclusion Criteria:

1) Adult patient booked for elective surgery requiring orotracheal intubation

Exclusion Criteria:

1. Any patient in whom the use of the GlideScope is contraindicated in the opinion of the attending anesthesiologist.
2. Any patient with cervical spine abnormalities.
3. Any patients with known or probable difficult airways.
4. Any patient requiring rapid sequence induction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of Intubation | During the intubation
  Duration of Intubation from mask removal to confirmation of ETCO2

SECONDARY OUTCOMES:
Ease of Intubation | Within 5 minutes of the completion of the intubation
  100 mm visual analog scale
Number of intubation attempts | Within 5 minutes of the completion of the intubation
  Number of intubation attempts
Failure to intubate | Within 5 minutes of the completion of the intubation
  Failure to intubate
Laryngoscopic Grade | Within 5 minutes of the completion of the intubation
  Cormack & Lehane grade
Oropharyngeal Trauma | Within 5 minutes of the completion of the intubation
  Blind suction of the oropharynx immediately post intubation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Turkstra, Principal Investigator — University of Western Ontario, Canada
Locations (2):
- Canada (2):
  - St. Joseph's Health Care, London, Ontario
  - London Health Sciences Center University Hospital, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turkstra TP, Turkstra DC, Pavlosky AW, Jones PM. Simultaneous en bloc endotracheal tube insertion with GlideScope(R) Titanium video laryngoscope use: a randomized-controlled trial. Can J Anaesth. 2020 Nov;67(11):1515-1523. doi: 10.1007/s12630-020-01778-2. Epub 2020 Aug 19. PMID 32815101